CLINICAL TRIAL: NCT06830356
Title: Somatostatin Receptor PET Imaging to Guide Radiotherapy Dose Escalation in High Risk Meningiomas.
Acronym: SPIDER-MEN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centro di Riferimento Oncologico - Aviano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRO-2024-47
Record Dates: First submitted 2025-02-11; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Meningioma
MeSH Terms: conditions — Meningioma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation of radiation therapy, based on somatostatin receptor PET imaging (Experimental): Radiation treatment with higher doses than the standard and defined using PET imaging
  Interventions: Radiation: Dose escalation of radiation therapy, based on somatostatin receptor PET imaging

INTERVENTIONS:
Radiation: Dose escalation of radiation therapy, based on somatostatin receptor PET imaging — Radiation treatment with higher doses than the standard and defined using PET imaging

SUMMARY:
High-risk meningiomas always require postsurgical radiation treatment. Recent evidence has shown that increased radiation therapy dose may be associated with increased intracranial control of disease. In order to better define the volume of radiation treatment, the addition of PET imaging with somatostatin receptor tracers adds additional information compared to encephalon MRI with MoC alone.The present study aims to investigate whether radiation treatment with higher doses than the standard and defined using PET imaging can be safe and at the same time effective in order to increase progression-free survival in high-risk meningiomas.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 16 years;
* Ability to express appropriate informed consent to treatment;
* Diagnosis of grade III meningioma (regardless of presence of residual) or diagnosis of recurrence of grade II meningioma (regardless of presence of residual) or first diagnosis of grade II meningioma with presence of residual;
* In case of recurrence, confirmation can be either histological or radiological;
* Not previous brain-level radiotherapy;
* Performance status: ECOG=0-2.

Exclusion Criteria:

* Refusal to radiation treatment (i.e., absence of signed informed consent);
* Other concomitant oncologic therapies
* Current pregnancy;
* Grade I meningiomas or Grade II meningiomas if operated on at first diagnosis with radical resection;
* Inability to perform MRI with MoC or PET.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2024-12-23 (Actual); Primary Completion 2037-12-23 (Estimated); Study Completion 2037-12-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of brain radionecrosis | up to 13 years
  Incidence of symptomatic brain radionecrosis (grade >=2 defined according to CTCAE scale v5.0).
Assess progression free survival (progression free survival = PFS) at 3 years | up to 13 years
  Percentage of patients alive and free of disease progression at 3 years after the start of radiotherapy (PFS rate). Progression will be defined as increase in size of treated lesions or appearance of new lesions (according to RANO meningioma criteria)

SECONDARY OUTCOMES:
Overall survival (Overall survival = OS) | up to 13 years
  Overall survival (OS) will be defined as time between enrollment and death
Incidence of other toxicities | up to 13 years
  Incidence of other neurological toxicities graded using the CTCAE scale v. 5.0
Concordance between GTV-RM and GTV-PET | up to 13 years
  Concordance will be measured according to Dice Similarity coefficient

CONTACTS AND LOCATIONS:
Overall Officials: Lorenzo Vinante, Principal Investigator — Centro di Riferimento Oncologico di Aviano (CRO)
Locations (1):
- Centro di Riferimento Oncologico di Aviano (CRO), Aviano, Pordenone, Italy